CLINICAL TRIAL: NCT02196675
Title: A Prospective, Multi-Center Evaluation of a Powered Surgical Stapler in Video-Assisted Thoracoscopic Lung Resection Procedures in Korea
Brief Title: Evaluation of a Powered Surgical Stapler in Video-Assisted Thoracoscopic Lung Resection Procedures in Korea
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC-13-003
Record Dates: First submitted 2014-07-19; First posted 2014-07-22 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-06

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VATS wedge resection or lobectomy: Single arm study Intervention: Device: Endocutter
  Interventions: Device: Endocutter

INTERVENTIONS:
Device: Endocutter — The study utilized Echelon FlexTM Powered ENDOPATH® Stapler (Ethicon, Cincinnati, USA) along with compatible cartridges: Gray (closed staple height, 0.75mm), White (1.0mm), Blue (1.5mm), Gold (1.8mm), Green (2.0mm), and Black (2.3mm).

SUMMARY:
Collection of real world outcomes of Video-Assisted Thoracoscopic Surgery (VATS) for lung cancer (lobectomy, wedge resection) using ECHELON FLEX™ Powered ENDOPATH® Staplers 45 mm and/or 60 mm (study devices) in a Korean population.

DETAILED DESCRIPTION:
This clinical trial assessed the use of a powered stapler for transection in VATS lung resection, where there is currently limited published clinical data. The primary study endpoint was occurrence and duration of air leak / prolonged air leak (PAL). Procedure details and perioperative outcomes associated with VATS lung resections were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed of NSCLC (up to and including Stage II), or individuals undergoing VATS diagnostic wedge resection in accordance with their institution's Standard of care (SOC);
* Scheduled for lung resection surgery (lobectomy or wedge resection) involving only one lobe of the lung;
* Performance status 0-1 (Eastern Cooperative Oncology Group classification);
* ASA score ≤ 3;
* No prior history of VATS or open lung surgery;
* Willing to give consent and comply with study-related evaluation and treatment schedule; and
* At least 19 years of age.

Exclusion Criteria:

* Active (subject currently receiving systemic treatment) bacterial infection or fungal infection;
* Systemic administration (intravenous or oral) of steroids, including herbal supplements that contain steroids, (within 30 days prior to study procedure);
* Chemotherapy or radiation therapy for lung cancer may not be performed for 30 days prior to the procedure;
* Scheduled concurrent surgical procedure other than wedge resection or lobectomy (central venous access - e.g., port placement, mediastinoscopy with lymph node sampling, and VATS lymphadenectomy are allowed);
* Pregnancy;
* Physical or psychological condition which would impair study participation;
* The patient is judged unsuitable for study participation by the Investigator for any other reason; or
* Unable or unwilling to attend follow-up visits and examinations.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with suspected or confirmed of NSCLC (up to and including Stage II), or individuals undergoing VATS diagnostic wedge resection in accordance with their institution's Standard of care (SOC);
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Fegelman, MD, Study Director — Johnson & Johson
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Samsung Medical Center, Seoul, Seoul
  - Asan Medical Center, Seoul, Seoul
  - Korean University Guro Hospital, Seoul, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals undergoing VATS lobectomy for suspected or confirmed Non-small Cell Lung Cancer, or individuals undergoing VATS diagnostic wedge resection in accordance with their institution's Standard of Care, and who meet study entry criteria, were enrolled in this study.
Pre-assignment Details: There was no assignment to treatment group given that this is a single arm study wherein the same device was used on all subjects. Results are presented for the overall cohort as well as by the individual procedure performed - lobectomy, wedge resection, or wedge resection with lobectomy.
Groups:
- Wedge Resection: Subjects undergoing VATS wedge resection using Echelon FlexTM Powered ENDOPATH® Stapler
- Lobectomy: Subjects undergoing VATS lobectomy using Echelon FlexTM Powered ENDOPATH® Stapler
- Wedge Resection With Lobectomy: Subjects undergoing VATS wedge resection that also required lobectomy using Echelon FlexTM Powered ENDOPATH® Stapler
Period: Overall Study
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Started | 27 | 70 | 8
Completed | 25 | 68 | 7
Not Completed | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Intra-operative surgical exclusion | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who consented to the study, had surgery for wedge resection, lobectomy, or wedge resection with lobectomy and were not converted to an open procedure. Two enrolled subjects were converted to an open procedure and thus were not included in this summary. These subjects were followed for safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy | Total
Number analyzed (Participants) | 26 | 69 | 8 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (11.39) | 60.5 (10.41) | 61.6 (8.09) | 61.2 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 31 | 5 | 49
  Male | 13 | 38 | 3 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 26 | 69 | 8 | 103
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 26 | 69 | 8 | 103

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Prolonged Air Leaks
Description: Prolonged air leaks defined as longer than 5 days in continuous duration. Air leak was to be quantitatively assessed starting on the evening after surgery and then twice daily (during morning and evening rounds). Patients were instructed to perform standardized repeated forced expiratory maneuvers (coughing and blowing).
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: All subjects who consented to the study, had surgery for wedge resection, lobectomy, or wedge resection with lobectomy and were not converted to an open procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Wedge Resection: Subjects undergoing VATS wedge resection
- Lobectomy: Subjects undergoing VATS lobectomy
- Wedge Resection With Lobectomy: Subjects undergoing VATS wedge resection that also required lobectomy
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 26 | 69 | 8
percentage of participants | 0.0 [0.0 to 13.2] | 5.8 [1.6 to 14.2] | 37.5 [8.5 to 75.5]

2. Secondary Outcome: Occurrence of Postoperative Air Leaks
Description: Air leak was to be quantitatively assessed starting on the evening after surgery and then twice daily (during morning and evening rounds). Patients were instructed to perform standardized repeated forced expiratory maneuvers (coughing and blowing).
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: ll subjects who consented to the study, had surgery for wedge resection, lobectomy, or wedge resection with lobectomy and were not converted to an open procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 26 | 69 | 8
percentage of participants | 30.8 [14.3 to 51.8] | 42.0 [30.2 to 54.5] | 75.0 [34.9 to 96.8]

3. Secondary Outcome: Length of Stay (LOS)
Description: Determined as the length of time in days from hospital admission to initial hospital discharge
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: All subjects who consented to the study, had surgery for wedge resection, lobectomy, or wedge resection with lobectomy and were not converted to an open procedure and had complete data. One subject was missing the hospital discharge date, thus length of stay could not be calculated.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 25 | 69 | 8
days | 7.2 (2.95) | 9.3 (4.07) | 9.4 (2.67)

4. Secondary Outcome: Volume of Estimated Intra-operative Blood Loss
Time Frame: Blood loss intra-op and up to 5 days post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 26 | 69 | 8
milliliters | 30.4 (40.27) | 146.1 (155.96) | 91.3 (124.95)

5. Secondary Outcome: Time to Chest Tube Removal
Description: Defined as the number of days from date of surgery to removal of the last chest tube inserted during the surgical procedure.
Time Frame: Post-operative period through hospital discharge and follow-up at Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Number analyzed (Participants) | 26 | 69 | 8
days | 3.4 (1.63) | 5.2 (1.97) | 6.3 (2.38)

ADVERSE EVENTS:
Time Frame: Duration of follow-up was scheduled through approximately 4 weeks post surgery
Arm/Group | Wedge Resection | Lobectomy | Wedge Resection With Lobectomy
Serious Adverse Events (participants affected / at risk) | 0/27 | 9/70 | 3/8
Other Adverse Events (participants affected / at risk) | 17/27 | 43/70 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wedge Resection (N=27) | Lobectomy (N=70) | Wedge Resection With Lobectomy (N=8)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Wedge Resection (N=27) | Lobectomy (N=70) | Wedge Resection With Lobectomy (N=8)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 17 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 12 | 15 | 1
Liver function test abnormal (Investigations) | 0 | 2 | 1
Dizziness (Nervous system disorders) | 4 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation, the Institution will provide Sponsor with at least sixty (60) days for review of a manuscript. Notwithstanding the foregoing, no paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written consent.